CLINICAL TRIAL: NCT06113653
Title: Outcomes and Predictors of Mortality Among Preterm Infants With Neonatal Sepsis Admitted in NICU of Assiut University Children's Hospital
Brief Title: Outcomes and Predictors of Mortality Among Preterm Infants With Neonatal Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmine Thabet Ragab, 71515assiut, Assiut University
Other Study IDs: Outcomes of neonatal sepsis
Record Dates: First submitted 2023-10-28; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis | interventions — Prospective Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prospective study — Prospective study of outcomes and predictors of mortality among preterm infants with neonatal sepsis

SUMMARY:
A prospective cross-sectional study of outcomes and predictors of mortality among preterm infants with neonatal sepsis admitted in NICU of Assiut University Children's Hospital

DETAILED DESCRIPTION:
Neonatal sepsis is a clinical syndrome of bacteremia with systemic signs and symptoms of infection in the first 28 days of life. It can also result from viral and fungal invasions of the bloodstream It is one of the events that can occur during neonatal intensive care unit (NICU) admission. It contributes significantly to the morbidity of very preterm (VP: <32 weeks gestational age) and/or very low birthweight (VLBW: <1500 g) infants Sepsis is a major cause of neonatal mortality and neurodevelopmental impairment among neonates which results in death and major disability for 39% of those affected even with timely antibiotic treatment .

Globally, it is estimated that more than 1.4 million neonatal deaths annually are the consequence of invasive infections .

Infection-specific mortality varies by geographic region and neonatal risk factors like gestational age and body weight .

It contributes to nearly 30-50% of neonatal deaths in developing countries . The risk of death is highest in the first 24 h of life when more than half of deaths occur and about three-quarters of all neonatal deaths occur within the first week of life.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants (<37 weeks) diagnosed with neonatal sepsis
* Preterm infants aged 0-28 days

Exclusion Criteria:

* Full term infants (> 37 weeks gestation) -Neonates with congenital anomalies -Neonates diagnosed with metabolic diseases
* Neonates with birth asphyxia

Ages: 1 Minute to 28 Days | Sex: All
Age Groups: Child
Study Population: All preterm infants diagnosed with neonatal sepsis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-28 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
mortality among preterm infants with neonatal sepsis | Baseline
  mortality among preterm infants with neonatal sepsis admitted in NICU of Assiut university children's hospital